CLINICAL TRIAL: NCT05613075
Title: Potential Effect Assessment of Locally Applied Hyaluronic Acid, When Mixed With Autogenous De-mineralized Tooth Graft, for Socket Preservation, in Comparison With the Application of Autogenous De-mineralized Tooth Graft Alone.
Brief Title: Effect of Hyaluronic Acid, With Demineralized Tooth Graft, in Socket Preservation, vs Demineralized Tooth Graft Alone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rahma Hesham Ahmed, dentistry post graduate master student, Implantology Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rahma.autograft
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Bone Resorption; Socket Preservation; Bone Resorption; Unrestorable Dentition
Keywords: dentin graft; autogenous tooth graft; socket preservation; hyaluronic acid
MeSH Terms: conditions — Bone Resorption | interventions — Tooth Extraction; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tooth extraction and socket preservation with demineralized tooth graft (Active Comparator): patients with immediate extraction sockets, filled and condensed with demineralized, autogenous dentinal graft particles, extracted and originated from the newly extracted tooth, then covered with biodegradable Gel foaming sponge.
  Interventions: Procedure: tooth extraction and socket preservation with demineralized tooth graft
- tooth extraction and socket preservation with demineralized tooth graft and hyaluronic acid (Experimental): patients with immediate extraction sockets, filled and condensed with demineralized, autogenous dentinal graft particles, extracted and originated from the newly extracted tooth, mixed with Hyaluronic acid, in gel form, as a carrier, then covered with biodegradable Gel foaming sponge.
  Interventions: Procedure: tooth extraction and socket preservation with demineralized tooth graft with hyaluronic acid

INTERVENTIONS:
Procedure: tooth extraction and socket preservation with demineralized tooth graft — tooth extraction and socket preservation with demineralized tooth graft
  Arms: tooth extraction and socket preservation with demineralized tooth graft
Procedure: tooth extraction and socket preservation with demineralized tooth graft with hyaluronic acid — tooth extraction and socket preservation with demineralized tooth graft with hyaluronic acid
  Arms: tooth extraction and socket preservation with demineralized tooth graft and hyaluronic acid

SUMMARY:
Many dentists, clinicians and researchers have conducted numerous trials, and put several materials and procedures under the test, in an attempt to preserve vertical and/or horizontal extraction sockets dimensions. The clinical consequences of post-extraction remodeling may affect the outcome of the ensuing therapies aimed at restoring the lost dentition, either by limiting the bone availability for ideal implant placement or by compromising the aesthetic result of the prosthetic restorations. In an attempt for ridge/socket preservation of a freshly extracted tooth socket/bed, this study aims to assess and compare between using autogenous tooth graft added with Hyaluronic acid, and the usage of the standardized autogenous tooth graft alone, regarding the potency, preservative feature, and quality of bone healing, density, and deposition. For a better restorative outcome using a delayed implant placement later on in the edentulous area.

DETAILED DESCRIPTION:
The available studies provide insufficient information to assess the efficacy of the usage of ha after tooth extraction in order to induce wound healing and accelerates bone deposition and differentiation. Hence, the purpose of this clinical trial is to investigate whether there is any beneficial value of local administration of 8% ha gel formulation (gengigel ®; farmalink saglik, istanbul, turkey) on the postoperative healing phase, bone density and ridge dimensions.

In an attempt for ridge/socket preservation of a freshly extracted tooth socket/bed, this study aims to assess and compare between using autogenous tooth graft added with Hyaluronic acid, and the usage of the standardized autogenous tooth graft alone, regarding the potency, preservative feature, and quality of bone healing, density, and deposition. For a better restorative outcome using a delayed implant placement later on in the e-dentulous area.

Our null hypothesis that post-extraction ridges preserved with Hyaluronic acid mixed with autogenous tooth grafts will present no significant higher bone density at extraction site, nor better dimensional preservation of the ridge tooth/teeth socket(s), vertically and/or horizontally, than the normalized/standardized ridge preservation using autogenous tooth graft particulates alone, carried to serve delayed implants placement later on, at extraction sites.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old or older.
* 2. Requiring alveolar preservation after tooth extraction prior to placement of dental implant.
* 3. Participants that are eligible for immediate implantation, yet having factors that are hindering these patients from immediate placement of an implant at the time of extraction (ex: Financial related factors - psychological factors - time related factors).
* 4. Motivated patients with good enough understanding of oral health measurements and importance.
* 5. Sufficient keratinized gingiva to cover the grafted bone. 6. The presence of dentition adjacent to the bone defect.
* 7. Patients who are healthy or have well-controlled systemic disease(s).
* 8. Teeth extractions are to be recommended due to trauma, caries, or periodontal diseases. * 9. Single rooted teeth from both arches.
* 10. No acute infections, pus formation, socket and bony discharges.
* 11. Hopeless teeth, to be extracted, are bounded both mesially and distally by adjacent, teeth.
* 12. Intact buccal bone of the teeth to be extracted.

Exclusion Criteria:

* 1. Heavy smokers (more than 10 cigarettes per day or an electronic cigarette dose of >6 mg/ml of nicotine).
* 2. Presence of active infection or severe inflammation in the intervention zone.
* 3. Relevant medical history that contraindicates implant surgery.
* 4. Immunosuppression (eg. Hiv, solid-organ transplants). 5. Head and neck-irradiated patients in the past 5 years. 6. Regular intake of bisphosphonates, anticoagulants, or anti-inflammatories.
* 7. Chronic drug abuse or alcoholic habits. 8. Patients with poor oral hygiene (full-mouth plaque score and full-mouth bleeding score >15%) and lack of motivation.
* 9. Uncontrolled diabetes (reported levels of glycated haemoglobin exceeding 7%).
* 10. Uncontrolled and /or untreated periodontal disease. 11. Patients who had previously received bone graft on the site to be operated. 12. Patients with significant comorbidity such as recent heart attack or coagulation disorder.
* 13. Pregnant subjects.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
(BLRW) | 6 months
  Bucco-lingual alveolar ridge width
(BRH) | 6 months
  Height of Buccal ridge
(LRH). | 6 months
  height of Lingual ridge

SECONDARY OUTCOMES:
Percentage of newly formed bone | 6 months
  percentage of newly formed lamellar bone bundles and/or newly formed bone trabeculae
soft tissue healing | 2 weeks
  percentage of complete post operative wound closure by soft tissues
residual graft | 6 months
  percentage of residual bone graft particles
Visual analogue score (VAS) | 2 weeks
  Patient's pain and discomfort, 0-10 score, 0 represents "no pain", 10 represents "as bad as possible"

CONTACTS AND LOCATIONS:
Overall Officials: Rahma H Mohamed Ali, Principal Investigator — Cairo University, Faculty of Dentistry
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Hesham R, Shemais N, Saleh HA, Fawzy El-Sayed K. Autogenous Demineralized Dentin Graft With High Molecular Weight Hyaluronic Acid in Ridge Preservation: Pilot Trial. Clin Implant Dent Relat Res. 2025 Dec;27(6):e70100. doi: 10.1111/cid.70100. PMID 41235610